CLINICAL TRIAL: NCT01164826
Title: A Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover Bioequivalence Study of Nabumetone 750 mg Tablets of Dr. Reddy's and Relafen® 750 mg Tablets of Glaxosmithkline, in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Nabumetone 750 mg Tablets of Dr. Reddy's Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. M.S. Mohan/ Vice President - R & D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-605/06-00
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Nabumetone
MeSH Terms: interventions — Nabumetone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nabumetone (Experimental): Nabumetone 750 mg Tablets of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Nabumetone
- Relafen (Active Comparator): Relafen® 750 mg Tablets of Glaxosmithkline Research Triangle Park, NC.
  Interventions: Drug: Relafen

INTERVENTIONS:
Drug: Nabumetone — Nabumetone 750 mg Tablets of Dr. Reddy's Laboratories Limited
  Other Names: Relafen® 750 mg Tablets
  Arms: Nabumetone
Drug: Relafen — Relafen® 750 mg Tablets of Glaxosmithkline Research Triangle Park, NC.
  Arms: Relafen

SUMMARY:
The purpose of this study is:

* To Assess the bioequivalence study of Nabumetone 750 mg tablets and Relafen® 750 mg tablets in healthy, adult, human subjects under fed conditions with a washout period of 16 days.
* To monitor adverse events and ensure the safety of subjects.

DETAILED DESCRIPTION:
A randomized, open label, two treatment, two period, two sequence, single dose crossover, bioequivalence study of nabumetone 750 mg tablets of Dr. Reddy's Laboratories Limited and Relafen® 750 mg tablets of Glaxosmithkline research triangle park, in healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

* Subjects who will provide written informed consent
* Subjects must be healthy human beings within 18-45 years of age (inclusive) weighing at least 50 kg.
* Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2
* Subjects must be of normal health, as determined by medical history and physical examination performed within 21 days prior to the commencement of the study.
* Subjects whose screening laboratory values are within normal limits or considered by the physician/investigator to be of no clinical significance.
* Have normal ECG, X-ray and vital signs.
* Availability of the subject for the entire study period and willingness to adhere to the protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

The subjects will be excluded based on the following criteria:

* Subjects incapable of understanding the informed consent.
* Subjects who have:

  1. Systolic blood pressure less than 90 mm of Hg and more than 140 mm of Hg
  2. Diastolic blood pressure less than 60 mm of Hg and more than 94 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the physician/investigator.
  3. Pulse rate below SO/min and above lOO/min.
* History of hypersensitivity or idiosyncratic reaction to Nabumetone or any other related drugs.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
* Clinically significant illness within 4 weeks before the start of the study.
* Consumption of grapefruit for the past ten days prior to the dosing day until the completion of the study.
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking from 48 hours before dosing and until the completion of the study.
* Subjects who has taken over the counter or prescribed medications for during the last7 days from the date of study.
* Subjects should not have taken enzyme modifying drugs or any systemic medication within the past 30 days prior to start of clinical study
* History of any psychiatric illness, which may impair the ability to provide written, informed consent.
* Subjects with clinically significant abnormal values of laboratory parameters.
* Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 330 rnL in the past 90 days before the date of start of study.
* Subjects with positive screen for drugs of abuse and alcohol.
* Any subject in whom Nabumetone is contraindicated for medical reasons.
* Any subject with recent history of surgery.
* A history of difficulty in donating blood.
* A positive hepatitis screen including hepatitis B surface antigen, anti HCV and Anti HAV antibodies
* A positive test result for HIV antibody and/or syphilis
* A recent history or presence of asthma (including aspirin induced asthma) or nasa polyp.
* A recent history of alcoholism < 2 years) or of moderate (180 mL/day) alcohol use,or consumption of alcohol within 48 hr prior to receiving Investigational Product.
* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the Investigational Product and throughout the subjects participation in the study. In any such case subject selection will be at the discretion of the Investigator / Medical expert.
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study is based on Cmax and AUC parameters | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mohan lal Siva Prasad Sayana, Principal Investigator — Bioserve Clinical Research Private Limited
Locations (1):
- Bioserve Clinical Research Pvt. Ltd., Hyderabad, Andhra Pradesh, India